CLINICAL TRIAL: NCT04343625
Title: Feasibility of a Modified Yoga Program to Improve Pain in an Assisted Living Facility
Brief Title: Feasibility Study of a Modified Yoga Program for Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: 5 Healthy Towns Foundation (Unknown)
Responsible Party: Principal Investigator, Cheryl LaMore, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00128999
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Depression, Anxiety; Fatigue; Pain, Chronic; Sleep
MeSH Terms: conditions — Depression; Anxiety Disorders; Fatigue; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified sitting, gentle yoga class (Experimental): Participants attended a modified sitting gentle yoga class,10 weekly classes, each 60 minutes in duration.
  Interventions: Behavioral: Modified yoga class

INTERVENTIONS:
Behavioral: Modified yoga class — Modified yoga was used to see if it would improve pain, fatigue, depression and anxiety, as well as improve sleep quality.

SUMMARY:
The purpose of this study is to determine whether a modified yoga program helps improve pain and function in elders age 65 years or older living in an assisted living community. Participation in regular physical activity, such as yoga, may improve strength and mobility and decrease pain. This study was developed to ascertain whether a modified yoga program improves pain and function in assisted-living elders, age 65 years and older.

DETAILED DESCRIPTION:
Chronic pain is costly and debilitating, affecting an estimated 100 million Americans and costing about $600 billion a year in indirect and direct medical costs. Managing chronic pain is difficult, requiring an array of pharmacologic and non-pharmacologic approaches to address not only pain, but relevant and intertwined domains of life such as sleep, energy, and mood. One such non-pharmacologic therapy is yoga. Systematic reviews of yoga clinical trials have shown that yoga is effective in managing low back and neck pain. However, these studies utilized younger populations, and no studies have characterized the effects of yoga for pain in the elderly. Given the rapidly growing aged population, the growing popularity of yoga, and the high prevalence of pain conditions among elderly individuals, studies that examine the effect of yoga on acute and chronic pain in the elderly are warranted. Thus the purpose of this proposal is to perform a pilot study to assess the feasibility and efficacy of yoga for managing chronic pain in elderly adults. This study will characterize whether such an intervention is feasible, assess whether a gentle yoga intervention improves subjective symptoms of pain, and investigate whether this yoga interventions decreases use of as needed pain relievers among elderly adults. This pilot study will characterize these effects in a sample of 60 elderly adults in at the United Methodist Retirement community in Chelsea, Michigan. The results of this study will be immediately translatable to members of this community in the short term, and nationwide in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Report chronic (>3months) clinically relevant pain, defined as a score of ≥3 on a 0-10 numeric pain scale, at least 3 of 7 days per week
* Must be current resident of the United Methodist Retirement Community or Silver Maples Assisted Living Community with medical record availability regarding medication use over the previous 10 weeks

Exclusion Criteria:

* Persons who have not lived at the facility long enough to analyze their medical records
* Having any medical condition or lack of physical capability that would prohibit safe participation in yoga exercise
* No regular yoga practice (regular yoga practice defined as ≥1 practice session/week)
* Cannot provide informed consent for study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 20 weeks
  The Brief Pain Inventory (BPI) is a 15-item self-report measure that has been validated for use in a wide variety of pain states. The BPI assesses for the presence of pain, pain intensity (i.e., worst, least, average, current) and functional interference from pain.

SECONDARY OUTCOMES:
Depression and anxiety as measured by The HADS scale | 20 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a brief 14-item instrument that will be used to classify individuals as having normal, mild, moderate, or severe levels of anxiety and depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl E LaMore, MD, Principal Investigator — University of Michigan
Locations (1):
- Dominos Farms, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No